CLINICAL TRIAL: NCT02530398
Title: Single-arm, Non-randomized, Open, Drug Tolerance Trial of Cinobufacini Injection Intraperitoneal Perfusion Treatment on Digestive System Cancer Patients With Ascites
Brief Title: A Tolerance Trial of Cinobufacini Injection Intraperitoneal Perfusion on Digestive System Cancer With Ascites
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Quanwang Li, Chief of oncology dept, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-XTCX-05
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Digestive System Cancer; Malignant Ascites
MeSH Terms: conditions — Digestive System Neoplasms | interventions — huachansu

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cinobufacini group (Experimental): 48 patients(half males and half females) will be in the group.Central venous catheters will be preserved for drainage of ascites, after the drainage of most of ascites, we will slowly inject a dilute concentration of cinobufacini injection with escalated dosage through the catheters. Then we will evaluate the observation indexes, including adverse events, vital signs, electrocardiogram, blood routine, urine routine, hepatic and renal function, etc.
  Interventions: Drug: Cinobufacini Injection

INTERVENTIONS:
Drug: Cinobufacini Injection — Cinobufacini injection is extracted from a traditional Chinese medicine Bufo toad skins, it's something cold and poisonous with damp evil. On one hand it can kill the cancer cells direct; on the other hand it has the ability to contract blood vessels and inhibit the formation of tumor new vessels. It has been widely used in the treatment of various malignancies.

SUMMARY:
To evaluate the tolerance and safety of cinobufacini injection intraperitoneal treatment on digestive system cancer patients with malignant ascites, and propose dosage regimens for future clinical trials. The clinical trial is divided into two parts, including single and successive administration.

DETAILED DESCRIPTION:
To evaluate the tolerance and safety of cinobufacini injection intraperitoneal treatment on digestive system cancer patients with malignant ascites, and propose dosage regimens for future clinical trials. A single-arm, non-randomized, open, drug tolerance trial will be conducted. The clinical trial is divided into two parts, including single and successive administration.The single administration includes 7 groups, dose is escalated from 15ml to 180ml, with 2-6 patients per dose level. Central venous catheters will be preserved for drainage of ascites, after the drainage of most of ascites, we will slowly inject a dilute concentration of cinobufacini injection with escalated dosage through the catheters. This treatment will be given only once, and the volunteers will be observed for 24 hours. Then we will evaluate the observation indexes, including adverse events, vital signs, electrocardiogram, blood routine, urine routine, hepatic and renal function, etc. The successive administration includes 2 groups, according to the result of single administration, choose the second largest tolerance dose to conduct the 1st group of successive administration. If there are significant adverse effects, then drop to a lower dose to conduct the 2nd group; if the trial shows no adverse effects, it upgrades to a higher dose (the maximum tolerated dose) to conduct the 2nd group. The treatment will be given 3 times a week, 2 weeks as a period. Adverse effects will be evaluated during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. digestive system cancer with malignant ascites;
2. the age of 18-80 years;
3. neither systemic chemotherapy, nor peritoneal perfusion therapy in 2 weeks;
4. no cinobufotalin preparations in 2 weeks;
5. ECOG score 0-3;
6. the amount of ascites is above level II (1000-3000ml);
7. volunteer to participate and sign informed consent.

Exclusion Criteria:

1. non-cancer causes of ascites, such as peritonitis, cirrhosis，hypoalbuminemia;
2. Had an allergy history to toad's skin or its products or had adverse reactions like arrhythmia when applied before;
3. B ultrasound or CT confirmed the peritoneal cavity is separated which will affect the treatment of ascites and the estimation of ascites;
4. The conditions admit and the patients would better to undergo chemotherapy of malignant ascites;
5. cardiac function is Ⅲ-Ⅳ;
6. ALT> 3 times upper limit and / or TBIL> 2 times upper limit;
7. renal function is phase 3 and above 3;
8. have severe neutropenia of degree II or above, and / or moderate or severe anemia, and / or thrombocytopenia of degree II or above;
9. Consolidated mental disorders.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
the grade of adverse events | 14 days
  According to The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE 4.0)，grade the severity of adverse events (AE) that occur with drug treatment，which include symptoms, electrocardiogram, blood routine, urine routine, hepatic and renal function. Each item is graded 1-5.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology dept; Dongfang Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China